**Protocol Title:** Socioecological Factors Associated with Ethnic Disparities in Bariatric Surgery

Utilization and Post-Operative Weight Loss (Substudy)

**Principal Investigator:** Benjamin Schneider, M.D.,

**Population:** A subgroup of 100 adults 18-60 years old, with a BMI >35 kg/m<sup>2</sup> or who have

had a weight loss surgery 8 months prior to enrollment will be invited to

participate in this substudy.

Number of Sites: UT Southwestern

Study Duration: 2 years

**Subject Duration:** Approximately 1-2 weeks (cross-sectional)

#### **General Information**

The prevalence of severe obesity has increased steadily in the United States population with ethnic minority groups being disproportionately affected. This study will allow the investigators to examine potential relationships between the blood and gut microbiotas of patients with obesity before and after weight loss surgery (WLS) and evaluate potential ethnic differences in the blood and gut microbiotas before and after the WLS.

### **Background Information**

- WLS has become not only an increasingly utilized obesity treatment option when conventional lifestyle change methods (decreased caloric intake, increased activity levels) fail, but also a safe and medically effective treatment choice for severe obesity (body mass index [BMI] > 40 kg/m2 or > 35 kg/m2 with > 1 comorbidity),<sup>1-6</sup> type 2 diabetes<sup>7-15</sup> and other cardiometabolic risk factors.<sup>16-27</sup> In fact, a large body of evidence including 11 randomized clinical trials<sup>28</sup> indicate that WLS is a highly effective procedure that can also reduce blood sugar levels below diabetic thresholds. Based on this strong evidence, a Joint Statement endorsed by 45 professional organizations, diabetes clinicians and researchers recommend that WLS be a standardized treatment option for people with diabetes, including those who are mildly obese and fail to respond to conventional treatment.<sup>28</sup> Moreover, obese individuals who undergo WLS live higher quality and longer lives than those who do not undergo the procedure.<sup>29-31</sup>
- In the UT Southwestern WLS program, where approximately 400 surgeries are completed per year (> 6,000 since 2001; 60% Hispanic, 25% NHB, 5-10% multiracial, 5% NHW, 80% women), only 45-50% of the medically-referred patients who attend an initial education seminar complete WLS within a 12-15 month period. (NHB Non-Hispanic Black; NHW Non-Hispanic White)

Findings from our research group show a lower post-operative weight loss in non-Hispanic Blacks than non-Hispanic Whites and Hispanics.<sup>37</sup> Reasons for the ethnic group disparities in post-WLS weight loss and comorbidity resolution are largely unknown.<sup>39-41</sup> Gut microbial composition could mediate, at least in part the discrepancies in the weight loss observed after WLS.<sup>42-48</sup> Specifically, NHB individuals experience significantly less post-surgery weight loss and diabetes-related improvement versus NHW.

In addition to gut microbial ethnic discrepancies, blood microbial differences could also be playing a factor in modulating the degree of weight loss or metabolic improvement post-surgery, however, no studies to this day have analyzed potential ethnic differences in blood microbial composition. Historically, blood has been considered as sterile and microbes were presumed to be only present in infections; however, bacteria have been shown to exist in the blood of healthy humans. One hypothesis that explains the presence of blood bacteria is the translocation of gut bacteria into the circulatory system. Such dysbiosis, previous infections, and other inflammatory conditions increase gut permeability to bacteria by creating dysfunction in the intestinal epithelial barrier. These mechanisms may explain the presence of blood bacteria in healthy individuals. Blood bacterial composition differs in people with infectious, sastrointestinal; Alack discretional; Cardiorespiratory; Alack discretional composition differs in people with infectious, sastrointestinal; Cardiorespiratory; Alack discretional disc

Both blood and gut microbiotas have been related to the degree of fat mass loss and metabolic improvement after WLS.<sup>72-78</sup> Thus, it is possible that both microbiomes may afford a valuable source of novel biomarkers and targets for therapeutic modulation for this patient population. Considering that the gut microbiota could be the origin of the bacterial species present in the blood, it is important to investigate the relationship between the blood and gut microbial composition and how it is affected by WLS and ethnicity. Considering the above, we propose the following aims:

## **Substudy Objectives:**

- AIM 1. Compare the relationship between the blood and the gut microbiomes among a sample of (1) pre-WLS and (2) 6-month post-WLS participants.
- Hypothesis<sub>1</sub>: Blood bacterial composition will resemble that of the gut microbiome among pre-WLS participants. Because the effect of WLS on the blood microbiome is not known, our post-WLS results will be mostly exploratory.
- AIM 2. Determine racial differences in the blood microbiome of the pre- and post-WLS groups.
- Hypothesis<sub>2</sub>: Ethnic differences will be detected in both the pre- and post-WLS groups.

### **Substudy Design**

- A subgroup of participants from the main study will be invited to participate in a cross-sectional substudy evaluating the relationship between blood and gut microbiotas. A total of 100 participants will be recruited, with an aim for 50 participants to be recruited from the "non-completers" and the other 50 participants to be recruited from the "6 months post-WLS" follow-up group of our main project.
- From each of these subgroups, the target is for 50% to be NHB and 50% to be NHW. This is, by the
  end of the study we will have 4 groups: (1) no-WLS NHB, (2) no-WLS NHW, (3) post-WLS NHB, and (4)
  post-WLS NHW.

## **Substudy Population**

- Inclusion criteria for substudy: Both groups will be 18-60 years old and will belong to either NHW or NHB ethnic groups. "No-WLS" participants will have a BMI >35 kg/m² (threshold BMI for WLS) whereas "6-8 months post-WLS" participants will have no BMI requirements.
- Exclusion criteria for substudy: having taken antibiotics in the previous 3 months; metformin, proton pump inhibitors, probiotics, or prebiotics in the previous month; currently following a vegetarian diet; pregnancy; having any infection in the previous month; having a comorbid disease that might alter the blood microbiome composition (e.g., renal failure) or the intestinal permeability (e.g., IBS); and having any electronic implants (e.g., pacemaker) or active prostheses.
- Recruitment Strategy for Substudy. By the time this IRB gets approved, all baseline samples from the main study would have already been collected. Therefore, we will recruit our non-surgery participants from the "non-completers" group from the main study. An email will be sent to all the participants that fall in this category and research spots will be provided on a first come first serve basis. Participants can e-consent online into the study. To recruit participants who have had bariatric surgery 6-8 months prior to their enrollment into the substudy, we will contact "early and late completers" who have already had the WLS but who have not done so more than 8 months ago. If additional participants are needed, particularly due to strict ethnic requirements (limited to NHW and NHB) we will first send invitation emails to the Weight Wellness Clinic patients, and if recruiting at the expected rate continues to be an issue we will advertise through IRB-approved flyers on social media or in the clinic setting.

# **Substudy Procedures**

- Nutrition. Before each stool sampling point, participants will be asked to record their dietary intake for the previous 3 days. This will allow us to determine whether participants' diets affect the outcome of interest.
- Body Weight. Participants will be weighed using a SECA body composition scale. Participants will come
  to the clinic/laboratory in fasting conditions (8-12h fast). Height and waist circumference (at both the
  maximum abdominal protuberance and the umbilicus) will also be collected.
- Blood Samples. Two tubes of blood samples (20 ml) will be collected per participant after a fasting period of 8-12 hours. The venipuncture site will be first cleaned with alcohol and the first aliquot of blood drawn will be used for regular blood analysis (to exclude any potential skin contamination of the specimen that might affect blood microbial analysis) whereas the second tube will be used for gut microbial analysis. The EDTA tube will measure glucose, insulin, lipopolysaccharides, and lipopolysaccharides binding protein. The second tube (a Zymo DNA/RNA Shield blood collection tube [Zymo Research, R1150]) will be used for blood microbial analysis. To prevent host contamination from obscuring microbial signatures, before 16S rRNA sequencing is done, blood DNA will be eliminated using a protocol that depletes host cells.
- Stool Samples. Participants will self-collect stool samples and will store them in Zymo DNA/RNA Shield fecal collection tubes (Zymo Research, R1101) in their homes. Participants will bring the samples to their blood sample collection visit. Stool DNA extraction and 16S rRNA sequencing will be performed on these samples.

16S rRNA Analysis. The hypervariable region V3 and V4 of the bacterial 16S rRNA gene will be captured using the Illumina Nextera protocol (Part # 15044223 Rev. B; Illumina, San Diego, CA). A single amplicon of 460bp will be amplified using the 16S Forward 5'TCGTCGGCAGCGTCAGATGTGTATAAGAGACAGCCTACGGGNGGCWGCAG and 16S Reverse Primer = 5'GTCTCGTGGGCTCGGAGATGTGTATAAGAGACAGGACTACHVGGGTATCTAATCC, as described in the Illumina protocol. A subset of samples n= 50) will be analyzed using a whole-genome metagenomic sequencing approach to validate 16S data as well as to predict and explore the genes and potential functional aspects of detected microbiota. The polymerase chain reaction (PCR) product will be cleaned using Agencourt AMPure XP beads (Agencourt Bioscience Corporation, A Beckman Coulter Company, Beverly, MA). The Illumina adapter and barcode sequences will be ligated to the PCR amplicons in order to attach them to a MiSeqDx flow cell for multiplexing. The quality and quantity of each sequencing library will be assessed using a bioanalyzer and PicoGreen (Molecular Probes, Inc., Eugene, OR) measurements, respectively. About 6pM of pooled library will be loaded onto a MiSeqDX flow cell and sequenced using a PE300 (Paired end 300 bp) v3 kit. Raw FASTQ files will be demultiplexed based on unique barcodes and assessed for quality. Samples with more than 50K QC pass sequencing reads will be used for downstream 16S OTU analysis. Taxonomic classification and Operational Taxonomic Unit (OTU) abundance analysis will be done using a CLC Bio Microbial Genomics Module (QIAGEN, Redwood City, CA). Individual sample reads will be annotated with the Greengenes database, and taxonomic features of the sample will be determined. Blood microbiome compositions will be compared pre- and post-intervention. Alpha and beta diversity analyses will be computed to understand the within-sample and between-samples diversity, respectively. Raw FASTQ files will be submitted to the Sequence Read Archive (SRA).

## **Compensation Substudy**

At the end of the substudy participants will receive a \$100 USD Amazon e-card in appreciation of their participation. The card will be mailed electronically to the previously provided e-mail address within a week of completion.

## **Data and Safety Monitoring**

All participants in the study will be evaluated for AEs from the time consent is signed through study completion or withdrawal. There are no anticipated adverse events for this study.

#### **Adverse Events**

For this study, an AE is defined as any untoward medical occurrence, unintended disease or injury or any untoward clinical signs in study subjects, that is related to study. The following adverse events are expected/anticipated and should not be recorded for the purpose of this study:

- •Discomfort at the site of blood draw
- Bruising, swelling, or bleeding around the site
- Lightheadedness/fainting
- •Mild infection at the site of blood draw

Conditions/diseases that are chronic but stable should not be recorded as adverse events. Any changes in a chronic condition of disease that are consistent with its natural progression are also not considered AEs and should not be recorded.

## **Serious Adverse Events**

Serious Adverse Events are defined as any event that results in death, is life-threatening, requires inpatient hospitalization or the prolongation of an existing hospitalization.

All adverse events will be monitored and tracked by the study team and/or Principal Investigator. These events will be recorded and reported via UTSW's HRPP Reporting Guidelines. The prevalence of adverse events, as needed, will be reported to UTSW IRB and NIH through annual reports.

All results of this trial will be reported yearly UT Southwestern's IRB. Trial procedures and progress as well as the occurrence of adverse events will be examined at 6-month intervals. Any action that results in the temporary or permanent suspension of the trial will be undertaken with consultation with the study's NIH project officer and the IRB.

### **Substudy Statistics**

To measure the overlap between blood and gut microbiomes we will use weighted Jaccard indices. To compare alpha diversities between groups, Wilcoxon rank test on previously individually calculated Shannon indices (phyloseq) will be utilized. PERMANOVA will be utilized to detect differentially abundance ASVs that represent OTUs in the bacterial genus or species level through DESeq2, edgeR, or metagenomicSeq. Por all analyses that involve multiple testing we will use the Benjamin Hochberg false discovery rate. Por all analyses that involve multiple testing we will use the Benjamin Hochberg false discovery rate.

#### **Ethics**

IRB approval will be sought from UT Southwestern under the UT System Reciprocity Agreement. For the sub-group, participants who have already been enrolled in our main study will be the first invited to participate. If additional participants are needed, they will be invited through the Weight Wellness Clinic at UT Southwestern and through IRB-approved flyers posted on social media.

#### Data handling and record-keeping

Quality control and assurance. Online data storage and management will be accomplished via a RedCap database. Regarding data/records confidentiality, we have an established set of procedures designed to ensure the protection of confidentiality. All records on study participants will be stored in locked file cabinets in the office of the research team, who will maintain strict control over these records. As in our other studies, we will use a record system in which all participant records are filed according to their assigned subject ID. Access to the database and data files is strictly controlled by the Principal Investigator. Passwords are used to restrict entry into the database. Project staff is specifically trained on issues of confidentiality. Facilitators will also be trained on issues of confidentiality.

Quality Assurance: Accuracy and Completeness of the Data During Data Collection, Entry, Transmission, and Analysis. The project TBA lead coordinator will be entrusted with scanning spot check 10% of the data after entry to ensure accuracy and check questionnaires for completeness as they are collected. Field team staff will follow-up with study participants concerning questions that are skipped. Participants are allowed to decline to answer but data checking is in place to ensure that data is not missing due to unintended circumstances.

**Data Integrity.** To maintain data integrity, fields within the RedCap database will have data type validation, simple ranges, and/or constraints. Data type validation will check that the entered data fits into the field type (i.e. a date field will only accept data entered in a date format). Simple ranges ensure that the data entered fits within the minimum and maximum values. Constraints check for invalid characters or values. Additionally more advanced checks can be done, such as cross-reference and

structured validations. Additionally, ad-hoc reports can be generated to check for data accuracy during the data collection process. Access to this feature will be restricted to required users using user privileges.

Data Export for Analysis. Data can be exported out from RedCap in various ways and in various formats. Data may be exported as a CSV (comma-delimited) file from a report or as a PDF file from the data entry page when viewing a particular record. Additionally, all collected data can be exported to CSV, XML, DBF, or Microsoft Excel file types. This interface allows for direct data importing, running SQL queries, generating ad-hoc reports, and accessing the data in real time. Access to these features will be restricted to authorized users using user privileges.

<u>Data Confidentiality</u>, <u>Storage and Preservation</u>. The PI and study team will have access for any required data cleaning. At the completion of the proposed study, access to database will be removed for all nonessential team members and further data modification will be disabled. All data will then be transferred from the database server into a 256-bit AES encrypted archive file and will only be accessible to the PI and a secondary co-custodian.

All participants will be assigned a unique code number by RedCap or the study team. This ID number will be used on all response forms, spreadsheets and data files to ensure participant confidentiality. Participant name, address, telephone, and any other means of identification will be destroyed following the completion of study using methods outlined by the UTSW HRPP office. All study personnel are equipped with password protected personal computer access and password protected access to a network drive accessible only from project staff computers. All computers and network drives are maintained by UT Health's Information Technology Department (IT).

<u>Data Security</u>. For added security and reliability, RedCap is separated into two servers, a web server and a database server. Data entry is done through the web server only and users do not have direct access to the database server. Both servers will be managed by UT Health's Information Technology and are physically located at its data center and covered by its security policies. Which include continuous network scans, penetration testing, daily patches, off-site tape backups, and other enterprise-level data management procedures. Additional security is implemented at the application level. RedCap maintains a built-in audit trail that logs all events, user access, and data creation and modifications. Log files can be exported for analysis and reporting purposes. All collected data is backed up hourly with redundant nightly backups stored to a separate server going back 6 months. Database consistency checks for errors and server maintenance also occur daily.

Finally, PI and the research team will meet regularly and follow appropriate compliance guidelines regarding data and safety.

#### **Publication Plan**

Results from this study will be published in leading peer-reviewed journals. Additionally, preliminary findings and analyses will be submitted to leading national and international research meetings in the field. The PI anticipates a minimum of 2 manuscripts published from the substudy. These aggregate results will be available to research subjects and they will be made aware of their existence.

#### **ATTACHMENTS**

- 1. Schematic of Study Design
- 2. Study Schedule
- 3. Consent Document

#### **References Cited:**

- 1. Flegal KM, Kruszon-Moran D, Carroll MD, Fryar CD, Ogden CL. Trends in Obesity Among Adults in the United States, 2005 to 2014. JAMA. 2016 Jun 7;315(21):2284-91.
- 2. Wang CY, Gortmaker SL, Taveras EM. Trends and racial/ethnic disparities in severe obesity among US children and adolescents, 1976-2006. Int J Pediatr Obes. 2011 Feb;6(1):12-20.
- 3. Karter AJ, Ferrara A, Liu JY, Moffet HH, Ackerson LM, Selby JV. Ethnic disparities indiabetic complications in an insured population. JAMA. 2002;287(19):2519-27.
- 4. McWilliams JM, Meara E, Zaslavsky AM, Ayanian JZ. Differences in control of cardiovascular disease and diabetes by race, ethnicity, and education: US trends from 1999 to 2006 and effects of Medicare coverage. Annals of Internal Medicine. 2009;150(8):505-15.
- 5. Zhang Q, Wang Y, Huang ES. Changes in racial/ethnic disparities in the prevalence of type 2 diabetes by obesity level among US adults. Ethnicity & Health. 2009;14(5):439-57.
- 6. Golden SH, Brown A, Cauley JA, Chin MH, Gary-Webb TL, Kim C, Sosa JA, Sumner AE, Anton B. Health disparities in endocrine disorders: biological, clinical, and nonclinical factors--an Endocrine Society scientific statement. J Clin Endocrinol Metab. 2012 Sep;97(9):E1579-639.
- 7. Pratt LA, Brody DJ. Depression and obesity in the U.S. adult household population, 2005- 2010.NCHS Data Brief. 2014 Oct;(167):1-8.
- 8. Sandoval JS, Harris JK, Jennings JP, Hinyard L, Banks G. Behavioral risk factors and Latino body mass index: a cross-sectional study in Missouri. J Health Care Poor Underserved. 2012 Nov;23(4):1750-67.
- Johnson NB, Hayes LD, Brown K, Hoo EC, Ethier KA. Centers for Disease Control and Prevention (CDC).
   CDC National Health Report: leading causes of morbidity and mortality and associated behavioral risk and protective factors--United States, 2005-2013. MMWR Surveill Summ. 2014 Oct 31;63 Suppl 4:3-27.
- 10. Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA 2004;292:1724–37.
- 11. Schauer PR, Kashyap SR, Wolski K, Brethauer SA, Navaneethan SD, Aminian A, Pothier CE, Kim ES, Nissen SE, Kashyap SR; STAMPEDE Investigators.. Bariatric surgery versus intensive medical therapy in obese patients with diabetes. N Engl J Med 2012;366:1567–76.
- 12. Sjöström L, Narbro K, Sjöström CD, Karason K, Larsson B, Wedel H, Lystig T, Sullivan M, Bouchard C, Carlsson B, Bengtsson C, Dahlgren S, Gummesson A, Jacobson P, Karlsson J, Lindroos AK, Lönroth H, Näslund I, Olbers T, Stenlöf K, Torgerson J, Agren G, Carlsson LM; Swedish Obese Subjects Study. Effects of bariatric surgery on mortality in Swedish obese subjects. N Engl J Med 2007;357:741–52.
- 13. Sugerman HJ, Starkey JV, Birkenhauer R. A randomized prospective trial of gastric bypass versus vertical banded gastroplasty for morbid obesity and their effects on sweets versus non-sweets eaters. Ann Surg 1987;205:613–24.
- 14. Schauer PR, Ikramuddin S, Gourash W, Ramanathan R, Luketich J. Outcomes afterlaparoscopic Roux-en-Y gastric bypass for morbid obesity. Ann Surg 2000;232:515–29.
- 15. Maggard MA, Shugarman LR, Suttorp M, Maglione M, Sugerman HJ, Livingston EH, Nguyen NT, Li Z, Mojica WA, Hilton L, Rhodes S, Morton SC, Shekelle PG. Meta-analysis: Surgical treatment of obesity. Ann Intern Med 2005;142:547–59.
- 16. Sjöström L, Lindroos AK, Peltonen M, Torgerson J, Bouchard C, Carlsson B, Dahlgren S, Larsson B, Narbro K, Sjöström CD, Sullivan M, Wedel H; Swedish Obese Subjects Study Scientific Group. Lifestyle, diabetes, and cardiovascular risk factors 10 years after bariatric surgery. N Engl J Med 2004;351:2683–93.
- 17. Dixon JB, O'Brien PE, Playfair J, J, Chapman L, Schachter LM, Skinner S, Proietto J, Bailey M, Anderson M. Adjustable gastric banding and conventional therapy for type 2 diabetes: a randomized controlled trial. JAMA 2008;299:316–23.
- 18. Mingrone G, Panunzi S, De Gaetano A, Guidone C, Raffaelli M, Callari C, Lombardi PC, Bellantone R. Bariatric surgery versus conventional medical therapy for type 2 diabetes. N Engl J Med 2012;366:1577–85.

- 19. Schauer PR, Kashyap SR, Wolski K, Wolski K, Brethauer SA, Navaneethan SD, Aminian A, Pothier CE, Kim ES, Nissen SE, Kashyap SR; STAMPEDE Investigators. Bariatric surgery versus intensive medical therapy in obese patients with diabetes. N Engl J Med 2012;366:1567–76.
- 20. De La Cruz-Munoz N, Messiah SE, Lopez-Mitnik G, Arheart KL, Lipshultz SE, Livingstone A. Laparoscopic Gastric Bypass Surgery and Adjustable Gastric Banding Significantly Decrease the Prevalence of Type 2 Diabetes Mellitus and Pre-Diabetes among Morbidly Obese Multiethnic Adults: Long-Term Outcome Results. J Amer Coll Surg 2011, Apr;212(4):505-11.
- 21. Buchwald H, Estok R, Fahrbach K, Banel D, Jensen MD, Pories WJ, Bantle JP, Sledge I. Weight and Type 2 Diabetes after Bariatric Surgery: Systematic Review and Meta-analysis. Am J Med 2009;122:248–56.
- 22. Shukla AP, Moreira M, Dakin G, Pomp A, Brillon D, Sinha N, Strain GW, Lebovitz H, Rubino F. Medical versus surgical treatment of type 2 diabetes: the search for level 1 evidence. Surg Obes Relat Dis 2012;8:476–82.
- 23. Sjöström L. Review of the key results from the Swedish Obese Subjects (SOS) trial—a prospective controlled intervention study of bariatric surgery. J Intern Med 2013;273:219–34.
- 24. Buchwald H, Varco RL, Matts JP, Long JM, Fitch LL, Campbell GS, Pearce MB, Yellin AE, Edmiston WA, Smink RD Jr, et al. Effect of partial ileal bypass surgery on mortality and morbidity from coronary heart disease in patients with Hypercholesterolemia: Report of the program on the surgical control of the Hyperlipidemias (POSCH). N Engl J Med 1990;323:946–55.
- 25. Christou NV, Sampalis JS, Liberman M, Look D, Auger S, McLean AP, MacLean LD. Surgery decreases long-term mortality, morbidity, and health care use in morbidly obese patients. Ann Surg 2004;240:416–24.
- 26. Adams TD, Gress RE, Smith SC, Halverson RC, Simper SC, Rosamond WD, Lamonte MJ, Stroup AM, Hunt SC. Long-term mortality after gastric bypass surgery. N Engl J Med 2007;357:753–61. Dixon JB, Bhathal PS, Hughes NR, O'Brien PE. Nonalcoholic fatty liver disease: improvement in liver histological analysis with weight loss. Hepatology 2004;39:1647–54.
- 27. Luyckx FH, Desaive C, Thiry A, Thiry A, Lefébvre PJ. Liver abnormalities in severely obese subjects: Effect of drastic weight loss after gastroplasty. Int J Obes 1998;22:222–6.
- 28. Rubino F, Nathan DM, Eckel RH, Schauer PR, Alberti KG, Zimmet PZ, Del Prato S, Ji L, Sadikot SM, Herman WH, Amiel SA, Kaplan LM, Taroncher-Oldenburg G, Cummings DE; Delegates of the 2nd Diabetes Surgery Summit.. Metabolic Surgery in the Treatment Algorithm for Type 2 Diabetes: a Joint Statement by International Diabetes Organizations. Obes Surg. 2017 Jan;27(1):2-21
- 29. Flum DR, Dellinger EP. Impact of gastric bypass operation on survival: Apopulation-based analysis. J Am Coll Surg 2004;199: 543–51.
- 30. Karlsson J, Sjöström L, Sullivan M. Swedish obese subjects (SOS) -An intervention study of obesity. Two-year follow-up of health related quality of life (HRQL) and eating behavior after gastric surgery for severe obesity. Int J Obes 1998;22:113–26.
- 31. Nguyen NT, Goldman C, Rosenquist CJ, Arango A, Cole CJ, Lee SJ, Wolfe BM. Laparoscopic versus open gastric bypass: a randomized study of outcomes, quality of life, and costs. Ann Surg 2001;234:279–91.
- 32. Buchwald H, Oien DM. Metabolic/bariatric surgery worldwide 2008. Obes Surg 2009;19:1605–11.
- 33. Pitzul KB, Jackson T, Crawford S, Kwong JC, Sockalingam S, Hawa R, Urbach D, Okrainec A. Understanding disposition after referral for bariatric surgery: when and why patients referred do not undergo surgery. Obes Surg. 2014 Jan;24(1):134-40.
- 34. Sadhasivam S, Larson CJ, Lambert PJ, Mathiason MA, Kothari SN. Refusals, denials, and patient choice: reasons prospective patients do not undergo bariatric surgery. Surg Obes Relat Dis. 2007 Sep-Oct;3(5):531-5.
- 35. Merrell J, Ashton K, Windover A, Heinberg L. Psychological risk may influence drop-out prior to bariatric surgery. Surg Obes Relat Dis. 2012 Jul-Aug;8(4):463-9.
- 36. Tsuda S, Barrios L, Schneider B, Jones DB. Factors affecting rejection of bariatric patients from an

- academic weight loss program. Surg Obes Relat Dis. 2009 Mar-Apr;5(2):199-202.
- 37. Khorgami Z, Arheart KL, Zhang C, Messiah SE, de la Cruz-Muñoz N. Effect of Ethnicity on Weight Loss After Bariatric Surgery. Obes Surg. May;25(5):769-76.
- 38. Khorgami Z, Zhang C, Messiah SE, de la Cruz-Muñoz N. Predictors of Post-Operative Aftercare Attrition among Gastric Bypass Patients. Bariatric Surgical Practice and Patient Care, 2015 Jun 1;10(2):79-83.
- 39. Lewis KH, Edwards-Hampton SA, Ard JD. Disparities in Treatment Uptake and Outcomes of Patients with Obesity in the USA. Curr Obes Rep. 2016 Jun;5(2):282-90.
- 40. Miller-Matero LR, Tobin ET, Clark S, Eshelman A, Genaw J. Pursuing bariatric surgery in an urban area: Gender and racial disparities and risk for psychiatric symptoms. Obesity Research and Clinical Practice 2016;10(1): 56–62.
- 41. Ortiz SE, Kawachi I, Boyce AM. The medicalization of obesity, bariatric surgery, and population health. Health (London). 2016 Aug 16. pii: 1363459316660858. [Epub ahead of print]
- 42. Chakaroun RM, Massier L, Heintz-Buschart A, et al. Circulating bacterial signature is linked to metabolic disease and shifts with metabolic alleviation after bariatric surgery. *Genome Med.* Jun 22 2021;13(1):105. doi:10.1186/s13073-021-00919-6
- 43. Murphy R, Tsai P, Jullig M, Liu A, Plank L, Booth M. Differential Changes in Gut Microbiota After Gastric Bypass and Sleeve Gastrectomy Bariatric Surgery Vary According to Diabetes Remission. *Obes Surg.* Apr 2017;27(4):917-925. doi:10.1007/s11695-016-2399-2
- 44. Al Assal K, Prifti E, Belda E, et al. Gut Microbiota Profile of Obese Diabetic Women Submitted to Rouxen-Y Gastric Bypass and Its Association with Food Intake and Postoperative Diabetes Remission. *Nutrients*. Jan 21 2020;12(2)doi:10.3390/nu12020278
- 45. Furet JP, Kong LC, Tap J, et al. Differential adaptation of human gut microbiota to bariatric surgery-induced weight loss: links with metabolic and low-grade inflammation markers. *Diabetes*. Dec 2010;59(12):3049-57. doi:10.2337/db10-0253
- 46. Graessler J, Qin Y, Zhong H, et al. Metagenomic sequencing of the human gut microbiome before and after bariatric surgery in obese patients with type 2 diabetes: correlation with inflammatory and metabolic parameters. *Pharmacogenomics J.* Dec 2013;13(6):514-22. doi:10.1038/tpj.2012.43
- 47. Wang FG, Bai RX, Yan WM, Yan M, Dong LY, Song MM. Differential composition of gut microbiota among healthy volunteers, morbidly obese patients and post-bariatric surgery patients. *Exp Ther Med*. Mar 2019;17(3):2268-2278. doi:10.3892/etm.2019.7200
- 48. Damms-Machado A, Mitra S, Schollenberger AE, et al. Effects of surgical and dietary weight loss therapy for obesity on gut microbiota composition
- 49. Brooks AW, Priya S, Blekhman R, Bordenstein SR. Gut microbiota diversity across ethnicities in the United States. *PLoS Biol*. Dec 2018;16(12):e2006842. doi:10.1371/journal.pbio.2006842
- 50. Nikkari S, McLaughlin IJ, Bi W, Dodge DE, Relman DA. Does blood of healthy subjects contain bacterial ribosomal DNA? *Journal of clinical microbiology*. May 2001;39(5):1956-9. doi:10.1128/JCM.39.5.1956-1959.2001
- 51. Paisse S, Valle C, Servant F, et al. Comprehensive description of blood microbiome from healthy donors assessed by 16S targeted metagenomic sequencing. *Transfusion*. May 2016;56(5):1138-47. doi:10.1111/trf.13477
- 52. Moriyama K, Ando C, Tashiro K, et al. Polymerase chain reaction detection of bacterial 16S rRNA gene in human blood. *Microbiol Immunol*. Jul 2008;52(7):375-82. doi:10.1111/j.1348-0421.2008.00048.x
- 53. McLaughlin RW, Vali H, Lau PC, et al. Are there naturally occurring pleomorphic bacteria in the blood of healthy humans? *Journal of clinical microbiology*. Dec 2002;40(12):4771-5. doi:10.1128/jcm.40.12.4771-4775.2002
- 54. Potgieter M, Bester J, Kell DB, Pretorius E. The dormant blood microbiome in chronic, inflammatory diseases. *FEMS Microbiol Rev.* Jul 2015;39(4):567-91. doi:10.1093/femsre/fuv013

- 55. Pretorius L, Kell DB, Pretorius E. Iron Dysregulation and Dormant Microbes as Causative Agents for Impaired Blood Rheology and Pathological Clotting in Alzheimer's Type Dementia. *Front Neurosci*. 2018;12:851. doi:10.3389/fnins.2018.00851
- 56. Pretorius L, Kell DB, Pretorius E. Iron Dysregulation and Dormant Microbes as Causative Agents for Impaired Blood Rheology and Pathological Clotting in Alzheimer's Type Dementia. *Front Neurosci*. 2018;12:851. doi:10.3389/fnins.2018.00851
- 57. Kell DB, Pretorius E. On the translocation of bacteria and their lipopolysaccharides between blood and peripheral locations in chronic, inflammatory diseases: the central roles of LPS and LPS-induced cell death. *Integr Biol (Camb)*. Nov 2015;7(11):1339-77. doi:10.1039/c5ib00158g
- 58. Castillo DJ, Rifkin RF, Cowan DA, Potgieter M. The Healthy Human Blood Microbiome: Fact or Fiction? *Front Cell Infect Microbiol*. 2019;9:148. doi:10.3389/fcimb.2019.00148
- 59. Li Q, Wang C, Tang C, Zhao X, He Q, Li J. Identification and Characterization of Blood and Neutrophil-Associated Microbiomes in Patients with Severe Acute Pancreatitis Using Next-Generation Sequencing. *Front Cell Infect Microbiol*. 2018;8:5. doi:10.3389/fcimb.2018.00005
- 60. Zrodlowski T, Sobonska J, Salamon D, McFarlane IM, Zietkiewicz M, Gosiewski T. Classical Microbiological Diagnostics of Bacteremia: Are the Negative Results Really Negative? What is the Laboratory Result Telling Us About the "Gold Standard"? *Microorganisms*. Feb 29 2020;8(3)doi:10.3390/microorganisms8030346
- 61. Puri P, Liangpunsakul S, Christensen JE, et al. The circulating microbiome signature and inferred functional metagenomics in alcoholic hepatitis. *Hepatology*. Apr 2018;67(4):1284-1302. doi:10.1002/hep.29623
- 62. Cho EJ, Leem S, Kim SA, et al. Circulating Microbiota-Based Metagenomic Signature for Detection of Hepatocellular Carcinoma. *Scientific reports*. May 17 2019;9(1):7536. doi:10.1038/s41598-019-44012-w
- 63. Dong Z, Chen B, Pan H, et al. Detection of Microbial 16S rRNA Gene in the Serum of Patients With Gastric Cancer. *Front Oncol.* 2019;9:608. doi:10.3389/fonc.2019.00608
- 64. Amar J, Lelouvier B, Servant F, et al. Blood Microbiota Modification After Myocardial Infarction Depends Upon Low-Density Lipoprotein Cholesterol Levels. *J Am Heart Assoc*. Oct 2019;8(19):e011797. doi:10.1161/JAHA.118.011797
- 65. Whittle E, Leonard MO, Harrison R, Gant TW, Tonge DP. Multi-Method Characterization of the Human Circulating Microbiome. *Front Microbiol*. 2018;9:3266. doi:10.3389/fmicb.2018.03266
- 66. Whittle E, Leonard MO, Gant TW, Tonge DP. Multi-Method Molecular Characterisation of Human Dust-Mite-associated Allergic Asthma. *Scientific reports*. Jun 20 2019;9(1):8912. doi:10.1038/s41598-019-45257-1
- 67. Qiu J, Zhou H, Jing Y, Dong C. Association between blood microbiome and type 2 diabetes mellitus: A nested case-control study. *J Clin Lab Anal*. May 2019;33(4):e22842. doi:10.1002/jcla.22842
- 68. Hammad DBM, Hider SL, Liyanapathirana VC, Tonge DP. Molecular Characterization of Circulating Microbiome Signatures in Rheumatoid Arthritis. *Front Cell Infect Microbiol*. 2019;9:440. doi:10.3389/fcimb.2019.00440
- 69. Bester J, Soma P, Kell DB, Pretorius E. Viscoelastic and ultrastructural characteristics of whole blood and plasma in Alzheimer-type dementia, and the possible role of bacterial lipopolysaccharides (LPS). *Oncotarget*. Nov 3 2015;6(34):35284-303. doi:10.18632/oncotarget.6074
- 70. Jin, Z., Chen, K., Zhou, Z. et al. Roux-en-Y gastric bypass potentially improved intestinal permeability by regulating gut innate immunity in diet-induced obese mice. Sci Rep 11, 14894 (2021). doi.org/10.1038/s41598-021-94094-8
- 71. James O'Brien, Denise Robertson, Bruce Griffin, Timothy Rockall, Chris Pring, EP.WE.824
  Effect of bariatric surgery on gut permeability in humans: a systematic review, British Journal of Surgery,
  Volume 108, Issue Supplement\_7, October 2021, znab308.095, doi.org/10.1093/bjs/znab308.095

- 72. Chakaroun RM, Massier L, Heintz-Buschart A, et al. Circulating bacterial signature is linked to metabolic disease and shifts with metabolic alleviation after bariatric surgery. *Genome Med.* Jun 22 2021;13(1):105. doi:10.1186/s13073-021-00919-6
- 73. Murphy R, Tsai P, Jullig M, Liu A, Plank L, Booth M. Differential Changes in Gut Microbiota After Gastric Bypass and Sleeve Gastrectomy Bariatric Surgery Vary According to Diabetes Remission. *Obes Surg.* Apr 2017;27(4):917-925. doi:10.1007/s11695-016-2399-2
- 74. Al Assal K, Prifti E, Belda E, et al. Gut Microbiota Profile of Obese Diabetic Women Submitted to Rouxen-Y Gastric Bypass and Its Association with Food Intake and Postoperative Diabetes Remission. *Nutrients*. Jan 21 2020;12(2)doi:10.3390/nu12020278
- 75. Furet JP, Kong LC, Tap J, et al. Differential adaptation of human gut microbiota to bariatric surgery-induced weight loss: links with metabolic and low-grade inflammation markers. *Diabetes*. Dec 2010;59(12):3049-57. doi:10.2337/db10-0253
- 76. Graessler J, Qin Y, Zhong H, et al. Metagenomic sequencing of the human gut microbiome before and after bariatric surgery in obese patients with type 2 diabetes: correlation with inflammatory and metabolic parameters. *Pharmacogenomics J*. Dec 2013;13(6):514-22. doi:10.1038/tpj.2012.43
- 77. Wang FG, Bai RX, Yan WM, Yan M, Dong LY, Song MM. Differential composition of gut microbiota among healthy volunteers, morbidly obese patients and post-bariatric surgery patients. *Exp Ther Med*. Mar 2019;17(3):2268-2278. doi:10.3892/etm.2019.7200
- 78. Damms-Machado A, Mitra S, Schollenberger AE, et al. Effects of surgical and dietary weight loss therapy for obesity on gut microbiota composition and nutrient absorption. *Biomed Res Int*. 2015;2015:806248. doi:10.1155/2015/806248
- 79. American Society for Metabolic and Bariatric Surgery and American College of Surgeons. Standards Manual V 2.0. Resources for optimal care of the metabolic and bariatric surgery patient 2016. Found at: https://www.facs.org/~/media/files/quality%20programs/bariatric/mbsaqip%20standardsmanual.ash x Accessed May 8, 2017.
- 80. Dreessen L, Arntz A Short-interval test-retest interrater reliability of the Structured Clinical Interview for DSM-III-R personality disorders (SCID-II) in outpatients. J Personal Disord 1998 Summer;12(2):138-48.
- 81. First MB, Spitzer RL, Gibbon M, Williams JBW, Davies M, Borus J, Howes MJ, Kane J, Pope HG, Rounsaville B. The Structured Clinical Interview for DSM-III-R Personality Disorders (SCID-II). Part II: Multi-site Test-retest Reliability Study, Journal of Personality Disorders 1995; 9(2), 92-104.
- 82. Fogelson DL, Neuchterlein KH, Asarnow RF, Subotnik KL, Talovic SA. Interrater Reliability of the Structured Clinical Interview for DSM-III-R, Axis II: Schizophrenia Spectrum and Affective Spectrum Disorders. Psychiatry Research 1991; 39:55-63.
- 83. Lobbestael J, Leurgans M, Arntz A. Inter-rater reliability of the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID I) and Axis II Disorders (SCID II). Clin Psychol Psychother 2011 Jan- Feb;18(1):75-9.
- 84. Maffei C, Fossati A, Agostoni I, Barraco A, Bagnato M, Deborah D, Namia C, Novella L, Petrachi M. Interrater reliability and internal consistency of the structured clinical interview for DSM-IV axis II personality disorders (SCID-II), version 2.0. J Personal Disord 1997 Fall;11(3):279-84.
- 85. Spadola CE, Wagner EF, Ruggianoa N; Accornero VH, E.; Vidot D, de la Cruz-Munoz N, Messiah SE. Urban, young adult bariatric surgery patients: Post-operative alcohol use, depression and anxiety. Accepted as a platform presentation to the 45th Annual Urban Affairs Association Conference, April 8- 11, 2015, Miami, FL
- 86. Walker SN, Sechrist KR, Pender NJ. The Health-Promoting Lifestyle Profile: Development and psychometric characteristics. Nursing Research 1987; 36(2):76-81.
- 87. Walker SN, Volkan K, Sechrist KR, Pender NJ. Health-promoting lifestyles of older adults: Comparisons with young and middle-aged adults, correlates and patterns. Advances in Nursing Science 1988; 11(1):76-90.
- 88. Walker, SN, Kerr MJ, Pender NJ, Sechrist KR. A Spanish language version of the Health Promoting

- Lifestyle Profile. Nursing Research 1990;39(5):268-273.
- 89. Dietary Screener Questionnaire in the NHANES 2009-2010. http://appliedresearch.cancer.gov/nhanes/dietscreen/
- 90. Gearhardt AN, Corbin WR, Brownell KD. Preliminary validation of the Yale Food AddictionScale. Appetite 2009; 52: 430-436.
- 91. Gearhardt AN, White MA, Masheb RM, Morgan PT, Crosby RD, Grilo, CM. An examination of the food addiction construct in obese patients with binge eating disorder. International Journal of Eating Disorders 2012; 45: 657-663.
- 92. Stunkard AJ, Messick S. The three-factor eating questionnaire to measure dietary restraint, disinhibition and hunger. Journal of Psychosomatic Research 1985;29(1):71-83.
- 93. Sallis JF, Kerr J, Carlson JA, Norman GJ, Saelens BE, Durant N, Ainsworth BE. Evaluating a brief self-report measure of neighborhood environments for physical activity research and surveillance: Physical activity neighborhood environment scale (PANES). Journal of Physical Activity and Health 2010; 7, 533-540.
- 94. http://www.cdc.gov/nchs/nhanes/nhanes2009-2010/PAQ\_F.htm
- 95. Moorehead MK, Ardelt-Gattinger E, Lechner H, Oria HE. The validation of the Moorehead-Ardelt Quality of Life Questionnaire II. Obes Surg. 2003 Oct;13(5):684-92.
- 96. Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. Journal of Health and Social Behavior 1983; 24:386-396.
- 97. Cohen S, Williamson G. Perceived Stress in a Probability Sample of the United States. Spacapan, S. and Oskamp, S. (Eds.) The Social Psychology of Health. Newbury Park, CA: Sage, 1988.
- 98. Rosenberg M, Schooler C, Schoenbach C, Rosenberg F. Global self-esteem and specific self- esteem. Amer Socio Rev 1995; 60: 141-56.
- 99. Avalos L, Tylka TL, Wood-Barcalow N. The Body Appreciation Scale: development and psychometric evaluation. Body Image. 2005 Sep;2(3):285-97.
- 100. Yang K, Zhang B, Kastanias P, Wang W, Okraniec A, Sockalingam S. Factors Leading to Self-Removal from the Bariatric Surgery Program After Attending the Orientation Session. Obes Surg. 2017 Jan;27(1):102-109.
- 101. Wharton S, Serodio KJ, Kuk JL, Sivapalan N, Craik A, Aarts MA. Interest, views and perceived barriers to bariatric surgery in patients with morbid obesity. Clin Obes. 2016 Apr;6(2):154-60.
- 102. Parma CD, Lee L, Sufi P. E-cigarette, obesity and Bariatric Surgery: Guidelines for the Bariatric Societies. Obesity surgery 2019; 29(9): 2982-2984.
- 103. Gorman-Smith D, Tolan PH, Zelli A, Huesmann R. The relation of family functioning to violence among inner-city minority youths. J. Fam. Psychol. 1996;10:115–129.
- 104. Tolan PH, Gorman-Smith D, Zelli A, Huesmann R. Assessment of family relationship characteristics: A measure to explain risk for antisocial behavior and depression among ur Canty- Mitchell, J. & Zimet, G.D. (2000). Psychometric properties of the Multidimensional Scale of Perceived Social Support in urban adolescents. American Journal of Community Psychology;28:391-400.
- 105. Zimet GD, Dahlem NW, Zimet SG, Farley GK. The Multidimensional Scale of Perceived Social Support. Journal of Personality Assessment 1988;52:30-41.
- 106. Zimet GD, Powell SS, Farley GK, Werkman S, Berkoff KA. Psychometric characteristics of the Multidimensional Scale of Perceived Social Support. Journal of Personality Assessment 1990;55:610-17.
- 107. Sallis JF, Grossman RM, Pinski RB, Patterson TL, Nader PR. The development of scales to measure social support for diet and exercise behaviors. Preventive Medicine 1987;16:825-836.
- 108. Stephenson M. Development and validation of the Stephenson Multigroup Acculturation Scale (SMAS). Psychol Assess. 2000 Mar;12(1):77-88.
- 109. Williams DR, Yu Y, Jackson JS, Anderson NB. Racial Differences in Physical and Mental Health: Socioeconomic Status, Stress, and Discrimination. Journal of Health Psychology. 1997; 2(3):335-351.
- 110. Taylor TR, Kamarck TW, Shiffman S. Validation of the Detroit area study discrimination scale in a

- community sample of older African American adults: the Pittsburgh healthy heart project. International Journal of Behavioral Medicine. 2004; 11:88–94.
- 111. Krieger N, Smith K, Naishadham D, Hartman C, Barbeau EM. Experiences of discrimination: validity and reliability of a self-report measure for population health research on racism and health. Social Science & Medicine. 2005; 61(7):1576-1596.
- 112. Marshall GN, Hays RD. The Patient Satisfaction Questionnaire Short Form (PSQ-18). Santa Monica, CA: RAND Corporation1994. p. 7865.
- 113. Poisson SN, Glidden D, Johnston SC, Fullerton HJ. Deaths from stroke in US young adults, 1989-2009. Neurology. 2014 Dec 2;83(23):2110-5.
- 114. Food Access Survey, Healthy Kids, Healthy Communities. Accessed March 20, 2015. Retrieved from:http://www.healthykidshealthycommunities.org/resources/neighborhood-food-access-survey
- 115. Spadola CE, Wagner EF, Ruggianoa N; Accornero VH, E.; Vidot D, de la Cruz-Munoz N, Messiah SE. Urban, young adult bariatric surgery patients: Post-operative alcohol use, depression and anxiety. Accepted as a platform presentation to the 45th Annual Urban Affairs Association Conference, April 8- 11, 2015, Miami, FL.
- 116. Vidot D, Prado G, Hlaing W, de la Cruz-Munoz N, Messiah SE. Relationship between Post- Operative Marijuana Use, Food Addiction, and Disordered Eating among Young Adult Bariatric Surgery Patients. Accepted as a poster presentation to the Scientific Sessions at the 31st Annual Meeting of the American Society for Metabolic and Bariatric Surgery at Obesity Week 2014, Nov. 2 7, 2014, Boston, MA
- 117. Centers for Disease Control and Prevention http://www.cdc.gov/healthyweight/assessing/bmi/adult\_bmi/index.html Accessed March 26, 2015.
- 118. http://www.metlife.com/Lifeadvice/Tools/Heightnweight/Docs/women.html
- 119. http://www.metlife.com/Lifeadvice/Tools/Heightnweight/Docs/men.html
- 120. http://www.metlife.com/Lifeadvice/Tools/Heightnweight/Docs/frametable.html
- 121. Huang TT, Johnson MS, Goran MI. Development of a prediction equation for insulin sensitivity from anthropometry and fasting insulin in prepubertal and early pubertal children: Diabetes Care. 2002 Jul;25(7):1203-10.
- 122. Public Health Service, Centers for Disease Control and Prevention. A proposed method for determining glucose using hexokinase and glucose-6-phosphate dehydrogenase. Center for Disease Control and Prevention,1-1-1976.
- 123. Allain CC, Poon LS, Chan CS, Richmond W, fu PC. Enzymatic determination of total serum cholesterol. Clin Chem 1974;20(4):470-475.
- 124. Burtis CA, Ashwood Er Border BP, Tietz NW. Tietz fundamentals of clinical chemistry. 5th ed ed. W.B. Saunders 2001.
- 125. Warnick GR, Mayfield C, Benderson J, Chen JS, Albers JJ. HDL-cholesterol quantitation by phosphotungstate-Mg2+ and by dextran sulfate-Mn2+-polyethylene glycol precipitation, both with enzymic cholesterol assay compared with the lipid research method. Am J Clin Pathol 1982; 78(5):718-723.
- 126. American Diabetes Association. Clinical practice recommendations 2002. Diabetes Care. 2002;25:S1-S147.
- 127. Simpson P, Gossett JM, Parker JG, Hall RA. Logistic regression modeling JMP start your analysis with a tree. Proceedings of the Twenty-Eighth Annual SAS Users Group International Conference 2003. Cary, NC: SAS Institute Inc. Available at: http://www2.sas.com/proceedings/sugi28/257-28.pdf.
- 128. Breiman L, Freidman JH, Olshen RA, Stone CJ. Classification and Regression Trees. Wadsworth: Belmont, CA, 1984.
- 129. Kiernan M, Kraemer HC, Winkleby MA, King AC, Taylor CB. Do logistic regression and signal detection identify different subgroups at risk? Implications for the design of tailored interventions. Psychological Methods 2001;6(1):35-48.

- 130. Westreich D, Lessler J, Funk MJ. Propensity score estimation: machine learning and classification methods as alternatives to logistic regression. Journal of Clinical Epidemiology 2010;63(8):826-833.
- 131. Swender H, Zucknick M, Ickstadt K, Bolt HM, A pilot study on the application of statistical classification procedures to molecular epidemiological data. Toxicology Letters 2004;151:291-299.
- 132. Gorroochurn P, Hodge SE, Heiman, GA, Durner M, Greenberg DA. Non-replication of association studies: pseudo failures to replicate. Genetics in Medicine 2007;9(6):325-331.
- 133. Nuzzo R. Statistical errors: P values, the gold standard of statistical validity are not as reliable as many scientist think. Nature 2014;506:150-152.
- 134. Breiman, L. Friedman, J., Olshen, R., and Stone, C. Classification and Regression Trees. Wadsworth International Group, Belmont, CA., 1984.
- 135. Kiernan, M., H. C. Kraemer, M. A. Winkleby, A. C. King, and C. B. Taylor. Do logistic regression and signal detection identify different subgroups at risk? Implications for the design of tailored interventions. Psychological Methods. 6:35-48, 2001.
- 136. Rakowski, W. and Clark, M.A. Do groups of women aged 50 to 75 match the national average mammography rate? American Journal of Preventive Medicine. 15(3):187-197, 1998.
- 137. Cook, N.R. Zee, R.Y.L. and Ridker, P.M. Tree and spline based association analysis of gene-gene interaction models for ischemic stroke. Statistics in Medicine. 24:1439-1453, 2004.
- 138. King, A.C. Kiernan, M. Oman, R.F. Kraemer H.C. Hull, M. Ahn, D. Can we identify who will adhere to long-term physical activity? Signal detection methodology as a potential aid to clinical decision making. Health Psychology. 16(4): 380-389.
- 139. Cohen, J. (1977). Statistical power analysis for the behavioral sciences (Revised Edition). New York, NY: Academic Press.
- 140. Ioannidis JPA. Why most published research findings are false. PLoS Medicine 2005;2(8):696-701.
- 141. McMurdie PJ, Holmes S. phyloseq: an R package for reproducible interactive analysis and graphics of microbiome census data. *PLoS One.* 2013;8(4):e61217.
- 142. Love MI, Huber W, Anders S. Moderated estimation of fold change and dispersion for RNA-seq data with DESeq2. *Genome biology*. 2014;15(12):550.
- 143. Robinson MD, McCarthy DJ, Smyth GK. edgeR: a Bioconductor package for differential expression analysis of digital gene expression data. *Bioinformatics*. 2010;26(1):139-140.
- 144. Paulson JN, Stine OC, Bravo HC, Pop M. Differential abundance analysis for microbial marker-gene surveys. *Nature methods.* 2013;10(12):1200-1202
- 145. Benjamini Y, Hochberg Y. Controlling the false discovery rate: a practical and powerful approach to multiple testing. *Journal of the royal statistical society Series B (Methodological)*. 1995:289-300
- 146. Essentials of Skeletal Radiology, 3rd ed, 2 vols. (2007). *Radiology, 243*(2), 348-348. doi: doi:10.1148/radiol.2432072509